CLINICAL TRIAL: NCT00492791
Title: Development and Validation of an Endoscopic Severity Score of Small Bowel Crohn's Disease With Wireless Capsule Endoscopy
Brief Title: Endoscopic Severity Score of Small Bowel Crohn's Disease With Wireless Capsule Endoscopy
Acronym: CAPSCDEIS
Status: Completed | Type: Observational
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Other Study IDs: GETAID 2006-2
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2011-08

CONDITIONS: Crohn's Disease
Keywords: crohn's disease; capsule endoscopes
MeSH Terms: conditions — Crohn Disease | interventions — Capsule Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic Capsule: Patient enrolled for performing an endoscopic capsule
  Interventions: Device: wireless endoscopy capsule

INTERVENTIONS:
Device: wireless endoscopy capsule — Firslty patency ingestion then wireless endoscopy capsule exam done

SUMMARY:
The endoscopic capsule is a new tool for exploration of the small intestine. The superiority of this technique on the radiological conventional examinations was shown in Crohn's disease. However no standardization of the lesions exists and no score of severity was proposed. The objective of this exploratory and multicentric study is to develop and validate an endoscopic score of severity especially dedicated to the examination by endoscopic capsule of the small intestine. Hundred twenty patients reached of disease of Crohn corresponding to various groups of severity will be included and will have an examination by video-capsule. The recorded examinations will be the standardized collection of all the lesions observed by independent readers, which will make it possible to evaluate the level of reproducibility of the detection of each lesion. Moreover, each reader will provide his total, qualitative and quantitative evaluations, of the severity of the attack of the small intestine. By using the data of only one reader, a score of severity will be built by simple linear function of the reproducible lesions observed. This score will be validated from the data corresponding to other readers of the same examinations, and those corresponding to another sample. Lastly, the aptitude of this score to detect the changes of the severity of the attack of the small intestine and to define the endoscopic cicatrization will be evaluated from data obtained among patients before and after treatment by infliximab or corticoids

DETAILED DESCRIPTION:
primary objective:Development and validation of an endoscopic score of severity of the small intestine adapted to its exploration by capsule among patients with crohn's disease secondary objectives:

* Study of the reproducibility of the detection of the lesions
* total evaluation of the severity of the small intestine (on an ordinal scale with 5 classes and on a continuous analogical scale).
* Study and validation of the sensitivity to the change of the score of severity (variation among patients after treatment by Infliximab or corticoids).
* Evaluation of the aptitude of the endoscopic score of severity to define the endoscopic cicatrization.
* Study of the correlation between the endoscopic score of severity and a clinical marker of activity: Crohn' S Disease Activity Index (CDAI) and a marker of inflammation: serum level of C-Reactive protein (CRP).
* Validation of the utility of "Patency Agile™" used before the capsule. All the patients included will have before their endoscopic capsule an examination by patency. After validation, the patients will have an exploration by the video capsule. The readers will fill a grid with standardized lesions. The films will be read by two other independent readers. The patients treated by infliximab or prednisone will have one second capsule afterwards 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Crohn's disease diagnosed on clinical, endoscopic, histological criteria. In active or inactive phase of their disease (HBI > 4; CDAI > 150).
* The patients will belong to the one of the 4 groups defined above according to the examinations carried out during the follow-up of the disease.
* Group 1: at least one ileal ulceration at ileocolonoscopy and no radiological abnormality
* Group 2: nonsevere attack on radiological examinations with or without endoscopic lesion
* Group 3: severe attack on radiological examinations with or without endoscopic lesion.
* Group 4: no lesion neither in endoscopy nor on radiologic exams.
* Small intestine standard exploration less than 1 year.
* Affiliation with the social security or a mode of social protection.
* able to understand and sign an informed consent.

Exclusion Criteria:

* ano-perineal location.
* Occlusion or sub-occlusion chronicle or intermittent or if there are frank signs of dilation of small intestine on the morphological examinations.
* Martial treatment since less than ten days before the realization of the capsule.
* Non steroidal anti-inflammatory treatment since less than three months before the realization of the capsule.
* Ileostomy on hail.
* Pace-maker or another implantable device.
* Swallowing troubles.
* Non evacuation of the Patency capsule in the 48 hours.
* Occlusion during the passage of the patency capsule.
* pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active or quiescent Crohn's Disease
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2007-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud BOURREILLE, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (20):
- Belgium (3):
  - Ulb - Clinique Saint Luc, Brussels
  - Gent University Hospital, Ghent
  - CHU LIEGE - Sart Tilman, Liège
- France (17):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - Hopital Saint Andre, Bordeaux
  - CHU CAEN, Caen
  - Hopital Beaujon, Clichy
  - Chru Lille, Lille
  - Chu Nantes, Nantes
  - CHU NICE, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Saint Louis, Paris
  - Hopital St Antoine, Paris
  - Hopital Georges Pompidou, Paris
  - Institut Mutualiste Montsouris (Imm), Paris
  - Chu Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - Chu Tours, Tours

REFERENCES:
- See also: Related Info — http://www.getaid.org/